CLINICAL TRIAL: NCT03590015
Title: Recruitment of Patients With Schizophrenia for "The Coronary Disease Project" Through Invitation Letters
Brief Title: Recruitment of Patients Through Invitation Letters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Bettina Ellen Grønbech, Research nurse, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Invitationsbrevet
Record Dates: First submitted 2018-07-06; First posted 2018-07-18 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Recruitment, Invitation Letters, Patients With Schizophrenia
Keywords: Recruitment; Invitation Letter; patients; Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- old letter of invitation (Other): Old invitation letter written by researchers/doctors in "The coronary project" sent to patients in order to recruit to an ongoing project
  Interventions: Other: Old invitation letter
- New letter of invitation (Other): New invitation Letter written with consideration of impaired language comprehension and has therefore been written in simple sentences with a sequential structure of basic information sent to patients in an ongoing project.
  Interventions: Other: New invitation Letter

INTERVENTIONS:
Other: Old invitation letter — Invitation Letter written by researchers/doctors
  Arms: old letter of invitation
Other: New invitation Letter — Invitation Letter written in simple sentences and a sequential structure of basic information in the rewritten information Letter
  Arms: New letter of invitation

SUMMARY:
Recruitment of patients with schizophrenia to clinical trials is difficult and in an ongoing project different methods of recruitment have been used in order to recruit. One of the methods used have been sending potential participant to the study an invitation letter with information of the study and an invitation to make contact with a project nurse. Not many patients have replied.

The aim of this study is to examine whether a simplified version of the invitation Letter, in terms of information structure and written style will encourage more patients to make contact to a project nurse.

DETAILED DESCRIPTION:
It is found that patients suffering from Schizophrenia have a positive attitude concerning participation in a research project but this doesn't always lead to recruitment. This might be due to schizophrenia being a disease causing self-disturbances in communication and contact to the surrounding World. It may lead to vulnerability in decision-making an a lower decision making capacity. Language disability is one of the most notable cognitive deficits in patients suffering from Schizophrenia and can be devided in to main components of usage and comprehension. Patients experience poorer listening comprehension and reading comprehension with no correlation to either age or education level and studies have shown that patients with schizophrenia have low literacy.

Therefore the aim of this study is to examine whether a rewritten version of an invitation Letter, taking in consideration patients low literacy and therefore written in simple sentences and with a sequential structure of information will make more patients take contact to a project nurse compared to patients receiving the original invitation Letter. The study design is a randomized controlled trial testing the old letter against the new letter.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Patients with a diagnosis within the spectre of Schizophrenia (F-20 to F-25) for at least ten years
* At the time of recruitment, a diagnosis of either F-20 or F-25 ( all diagnoses from ICD-10)
* Recidency in the Northern part of Jutland
* In treatment by an outpatient team
* Low frequency of contact with a clinician, once a month at the most

Exclusion Criteria:

* No exclusion criteria for receiving an invitation Letter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Response rates to the invitation Letters to be compared | within 3 weeks from receiving an invitation Letter
  response made to project nurse either by E-mail or phone

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Grønbech, nurse, Principal Investigator — Aalborg University Hospital
Locations (1):
- Bettina Ellen Grønbech, Aalborg, Northern Part of Jutland, Denmark